CLINICAL TRIAL: NCT03423940
Title: Basic and Clinical Studies in Reinforcing Positive Behaviors in Intellectual and Developmental Disabilities
Brief Title: Resurgence as Choice: Basic and Clinical Studies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Utah State University (Other)
Responsible Party: Principal Investigator, Brian D. Greer, Ph.D., BCBA-D, Consortium Principal Investigator, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro2019001815
Record Dates: First submitted 2018-01-19; First posted 2018-02-06 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-04

CONDITIONS: Problem Behavior; Self-injury; Communication
MeSH Terms: conditions — Problem Behavior; Self-Injurious Behavior; Communication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evaluation of Treatment Dosage (Experimental): In Arm 1, we will examine the optimal duration of treatment with functional communication training (FCT). Investigators will treat each participant's behavior using FCT in three distinct contexts which will be associated with either short, moderate, or extended treatment durations. The investigators will counterbalance the order of treatment durations (short, moderate, and extended) across participants, but each individual will receive treatment at each duration. Resurgence will be tested following each treatment duration.
  Interventions: Behavioral: Functional communication training
- Evaluation of Size of Decrease in Alternative Reinforcement (Experimental): In Arm 2, we will evaluate whether smaller, rather than larger, decreases in the availability of alternative reinforcement decreases the magnitude of resurgence. Investigators will counterbalance the order of differently sized decreases in alternative reinforcement with half of the participants in Arm 2 to determine whether the order of such decreases also affects resurgence magnitude.
  Interventions: Behavioral: Functional communication training

INTERVENTIONS:
Behavioral: Functional communication training — During functional communication training (FCT), the social consequence (e.g., attention, toys, breaks from instructions) that heretofore reinforced destructive behavior (i.e., as determined through a functional analysis) is delivered contingent on an appropriate communication response, while destructive behavior is on extinction (i.e., reinforcers are no longer provided). For example, if a functional analysis shows that aggression is reinforced by escape from demands, FCT would typically involve (a) teaching the child to access breaks from demands via a functional communication response (FCR; e.g., saying, "Break, please") and (b) placing destructive behavior on extinction (i.e., continuing with scheduled demands independent of destructive behavior).

SUMMARY:
Background: Functional communication training (FCT) is a commonly used intervention for teaching appropriate communication skills to children with intellectual disabilities who exhibit severe destructive behavior. Resurgence as Choice (RaC) Theory, a quantitative model of behavior, may help to explain why treatment relapse often occurs after FCT. This project will use the predictions of RaC to improve FCT treatments.

Objective: To test the predictions made by RaC with human participants who exhibit severe destructive behavior.

Eligibility: Children between the ages of 3 and 19 who display destructive behavior that is maintained by social consequences, who have IQ and adaptive behavior scores between 35 and 70, who are on a stable psychoactive drug regimen (or drug free) for at least 10 half-lives of each medication with no anticipated changes, and who have a stable educational plan and placement will be be eligible to enroll.

DETAILED DESCRIPTION:
Children with intellectual disabilities often display severe destructive behaviors that pose significant risk to self or others and represent barriers to community integration. These destructive behaviors are often treated with behavioral interventions derived from a functional analysis (FA), which is used to identify the environmental antecedents and consequences that occasion and reinforce (i.e., reward) the target response. One such treatment is called differential reinforcement of alternative behavior (DRA), which involves extinction (i.e., removal of rewards) of destructive behavior and reinforcement of an alternative communication response with the consequence that previously reinforced destructive behavior. Results from review studies indicate that interventions based on an FA, like DRA, typically reduce problem behavior by 90% or more.

One commonly used DRA intervention is functional communication training (FCT). During FCT, clinicians withhold reinforcement for destructive behavior and teach the individual a functional communication response to access reinforcement. For instance, a clinician may teach the child to exchange communication cards to express their wants and needs. However, DRA interventions reported in the literature have typically been evaluated by experts in controlled research settings, and treatment relapse often occurs in the natural environment when a caregiver is unable reinforce the DRA response every time that the response occurs due to competing responsibilities. Accordingly, a recent investigation of 25 applications of DRA found that relapse of problem behavior occurred in 76% of cases.

Resurgence as Choice Theory helps to explain why treatment relapse occurs under these circumstances and also provides mathematical equations that can be used to predict the variables that increase and decrease the likelihood that treatment relapse will occur. In this project, the investigators have used these equations to identify refinements to DRA that are likely to decrease the probability that treatment relapse will occur when the DRA response is not reinforced. In some cases, these refinements are at odds with what is recommended in the clinical literature on DRA. Therefore, it is important to evaluate these refinements that are derived from Resurgence as Choice Theory in order to determine the best way to implement DRA, so that treatment remains effective when it is implemented with less than perfect precision by caregivers in the natural environment.

The two predictions that are most relevant to our project are (a) resurgence of destructive behavior will decrease with increased DRA treatment duration, and (b) resurgence of destructive behavior will decrease with smaller, rather than larger, decreases in the availability of alternative reinforcement during the process of reinforcement schedule thinning. Accordingly, our project will examine the effects of different durations of DRA on resurgence and evaluate the effects of differently sized decreases in the availability of reinforcement to avoid resurgence. Findings from this project could have vast clinical implications for the treatment of severe destructive behavior.

ELIGIBILITY:
Inclusion Criteria:

1. males and females between the ages of 3 and 19;
2. problem behavior (e.g., aggression, property destruction, self-injurious behavior) that has been the focus of outpatient behavioral and pharmacological treatment but continues to occur, on average, more than once per hour;
3. problem behavior reinforced by social consequences (i.e., significantly higher and stable rates of the behavior in one or more social test conditions of a functional analysis [e.g., attention, escape] relative to the control condition [play] and the test condition for automatic reinforcement [alone or ignore]);
4. IQ and adaptive behavior scores between 35 and 70 (i.e., mild to moderate intellectual disability);
5. on a stable psychoactive drug regimen (or drug free) for at least 10 half-lives of each medication with no anticipated changes;
6. stable educational plan and placement, with no anticipated changes during the study.

Exclusion Criteria:

- Exclusion criteria.

1. children not meeting the inclusion criteria above;
2. children currently receiving intensive (i.e., 15 or more hours per week), function-based, behavioral treatment for their problem behavior through the school or another program;
3. DSM-V diagnosis of Rett syndrome or other degenerative conditions (e.g., inborn error of metabolism);
4. presence of a comorbid health condition (e.g., blindness) or major mental disorder (e.g., bipolar disorder) that would interfere with participation in the study (e.g., requiring frequent hospitalizations);
5. children with self-injurious behavior who, based on the results of the risk assessment, cannot be exposed to baseline conditions without placing them at risk of serious or permanent harm (e.g., detached retinas);
6. children requiring changes in drug treatment (but such children will be invited to participate after they meet the above criteria for a stable drug regimen).

Ages: 3 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-08-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers University Center for Autism Research, Education, and Services, Somerset, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share our outcome data using the National Database on Autism Research (NDAR). The investigators also plan to share our outcome data on the human participants in these two experiments who are not diagnosed with autism spectrum disorder to better understand how complex, comorbid disorders (e.g., self-injury) differ in individuals with and without autism spectrum disorder.

REFERENCES:
- [Background] Greer BD, Fisher WW, Saini V, Owen TM, Jones JK. Functional communication training during reinforcement schedule thinning: An analysis of 25 applications. J Appl Behav Anal. 2016 Mar;49(1):105-21. doi: 10.1002/jaba.265. Epub 2015 Oct 20. PMID 26482103
- [Background] Shahan TA, Craig AR. Resurgence as Choice. Behav Processes. 2017 Aug;141(Pt 1):100-127. doi: 10.1016/j.beproc.2016.10.006. Epub 2016 Oct 26. PMID 27794452
- [Background] Craig AR, Shahan TA. Behavioral momentum theory fails to account for the effects of reinforcement rate on resurgence. J Exp Anal Behav. 2016 May;105(3):375-92. doi: 10.1002/jeab.207. PMID 27193242
- [Background] Carr EG, Durand VM. Reducing behavior problems through functional communication training. J Appl Behav Anal. 1985 Summer;18(2):111-26. doi: 10.1901/jaba.1985.18-111. PMID 2410400
- [Background] Iwata BA, Dorsey MF, Slifer KJ, Bauman KE, Richman GS. Toward a functional analysis of self-injury. J Appl Behav Anal. 1994 Summer;27(2):197-209. doi: 10.1901/jaba.1994.27-197. PMID 8063622
- [Background] Tiger JH, Hanley GP, Bruzek J. Functional communication training: a review and practical guide. Behav Anal Pract. 2008 Spring;1(1):16-23. doi: 10.1007/BF03391716. PMID 22477675
- [Background] Shadish WR, Hedges LV, Pustejovsky JE. Analysis and meta-analysis of single-case designs with a standardized mean difference statistic: a primer and applications. J Sch Psychol. 2014 Apr;52(2):123-47. doi: 10.1016/j.jsp.2013.11.005. Epub 2013 Dec 27. PMID 24606972
- [Background] Hagopian LP, Boelter EW, Jarmolowicz DP. Reinforcement schedule thinning following functional communication training: review and recommendations. Behav Anal Pract. 2011 Summer;4(1):4-16. doi: 10.1007/BF03391770. PMID 22532899
- [Background] Saini V, Miller SA, Fisher WW. Multiple schedules in practical application: Research trends and implications for future investigation. J Appl Behav Anal. 2016 Jun;49(2):421-44. doi: 10.1002/jaba.300. Epub 2016 Mar 15. PMID 26990754
- [Background] Fisher WW, Kelley ME, Lomas JE. Visual aids and structured criteria for improving visual inspection and interpretation of single-case designs. J Appl Behav Anal. 2003 Fall;36(3):387-406. doi: 10.1901/jaba.2003.36-387. PMID 14596583
- [Background] Hyman SL, Fisher W, Mercugliano M, Cataldo MF. Children with self-injurious behavior. Pediatrics. 1990 Mar;85(3 Pt 2):437-41. PMID 2304806
- [Background] Emerson E, Kiernan C, Alborz A, Reeves D, Mason H, Swarbrick R, Mason L, Hatton C. The prevalence of challenging behaviors: a total population study. Res Dev Disabil. 2001 Jan-Feb;22(1):77-93. doi: 10.1016/s0891-4222(00)00061-5. PMID 11263632

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Evaluation of Treatment Dosage | Evaluation of Size of Decrease in Alternative Reinforcement
Started | 5 | 12
Completed | 4 | 9
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Evaluation of Treatment Dosage | Evaluation of Size of Decrease in Alternative Reinforcement | Total
Number analyzed (Participants) | 4 | 11 | 15
Age, Continuous [Mean (Full Range); unit: Years] | 8.75 [7 to 10] | 11.45 [4 to 19] | 10.73 [4 to 19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 4 | 9 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 2 | 6 | 8
  Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 6 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 5 | 7
Responses per minute of combined destructive behavior at or above 1.0 in baseline [Count of Participants; unit: Participants] — Combined destructive behavior (e.g., self-injury, aggression) will be at or above 1.0 responses per minute in baseline.
  Participants | 4 | 11 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Showing Resurgence as Predicted by the Quantitative Model -- Highest Response Rate
Description: Mean responses per minute of destructive during the resurgence test conditions are compared within-participant to determine whether response rates are highest in the test condition predicted by the model to produce the highest rate of responding.
Time Frame: Through study completion, an average of 4 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Evaluation of Treatment Dosage | Evaluation of Size of Decrease in Alternative Reinforcement
Number analyzed (Participants) | 3 | 9
Participants | 1 | 5

2. Secondary Outcome: Number of Participants Showing Resurgence as Predicted by the Quantitative Model -- Lowest Response Rate
Description: Mean responses per minute of destructive during the resurgence test conditions are compared within-participant to determine whether response rates are lowest in the test condition predicted by the model to produce the lowest rate of responding.
Time Frame: Through study completion, an average of 4 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Evaluation of Treatment Dosage | Evaluation of Size of Decrease in Alternative Reinforcement
Number analyzed (Participants) | 3 | 9
Participants | 2 | 6

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 4 months.
Arm/Group | Evaluation of Treatment Dosage | Evaluation of Size of Decrease in Alternative Reinforcement
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/11
Other Adverse Events (participants affected / at risk) | 0/4 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/40/NCT03423940/Prot_001.pdf
  • Statistical Analysis Plan (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/40/NCT03423940/SAP_002.pdf
  • Informed Consent Form (2023-05-03): https://cdn.clinicaltrials.gov/large-docs/40/NCT03423940/ICF_003.pdf